CLINICAL TRIAL: NCT03325244
Title: The Impact of Night Float on Anesthesiology Resident Sleep Patterns
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Lauren Dunn, MD, Assistant Professor of Anesthesiology, University of Virginia
Other Study IDs: 11590
Record Dates: First submitted 2017-04-07; First posted 2017-10-30 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All participants will use a portable EEG monitor and FITBIT to monitor sleep and activity before and after night call
  Interventions: Other: EEG monitor; Other: FitBit

INTERVENTIONS:
Other: EEG monitor — sleep patterns will be monitored using EEG monitor
Other: FitBit — activity levels will be monitored

SUMMARY:
Residency training requires hospital presence twenty-four hours a day. At times this necessitates working extended shifts, including night shifts, resulting in altered sleep patterns and sleep deprivation. Since 2003, the Accreditation Council for Graduate Medical Education (ACGME) has enforced duty hour regulations limiting shift length, the amount of weekly hours worked, and other variables governing shift work. Numerous studies have sought to determine the impact of duty hour regulations on the quality of patient care and resident education.

In addition to affecting patient care, medical resident sleep deprivation also has the potential to affect residents' well-being and their ability to perform basic tasks. A study in surgical residents showed reduced efficiency and safety in performing simulated laparoscopy following a period of sleep deprivation that was worse with novices compared to experienced residents. Recently, UVA found that resident physicians have greater difficulty controlling speed and driving performance with increased reaction times and minor and major lapses in attention in the driving simulator following six consecutive night shifts.

To comply with duty hour restrictions, residency programs have adopted various strategies including the creation of night float systems where residents are required to work multiple nights in a row. Reduced shift length has been associated with decreased medical errors, motor vehicle collisions, and percutaneous injuries.Surgical residents who transitioned to a night float system from 24-hour call every 3rd day reported reduced fatigue, more time for sleep and independent reading and increased family time, while nurses and patients reported improved communication and quality of patient care. In a pilot study of urology residents assigned to a 12-hour day shift (Monday-Friday), 12-hour night float (Sunday-Friday) or 24-hour home call, actigraphy was used to measure total sleep time, sleep latency and depth of sleep. Night float did not impact total sleep time or quality of sleep. However, these studies did not establish the optimal shift duration

DETAILED DESCRIPTION:
Participants wear a portable EEG monitor and a FITBIT activity monitor while attempting to sleep while on night call and at home for a baseline reading

ELIGIBILITY:
Inclusion Criteria:

* postgraduate year (PGY) 2, 3, and 4 Anesthesia residents

Exclusion Criteria:

* history of pacemaker or other medical device
* unable or unwilling to consent and comply with the protocol
* history of sleep disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postgraduate year (PGY) 2, 3, and 4 Anesthesia residents
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
sleep time | daily over 13 day period (Day 1 -Day 12)
  total sleep time as measured by EEG monitor

SECONDARY OUTCOMES:
activity level | daily over 13 day period (Day 1-Day 12)
  • as measured by activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Dunn, MD, Principal Investigator — University of Virginia Depaertment of Anesthesiolgy
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philibert I, Nasca T, Brigham T, Shapiro J. Duty-hour limits and patient care and resident outcomes: can high-quality studies offer insight into complex relationships? Annu Rev Med. 2013;64:467-83. doi: 10.1146/annurev-med-120711-135717. Epub 2012 Oct 26. PMID 23121182
- [Background] Sen S, Kranzler HR, Didwania AK, Schwartz AC, Amarnath S, Kolars JC, Dalack GW, Nichols B, Guille C. Effects of the 2011 duty hour reforms on interns and their patients: a prospective longitudinal cohort study. JAMA Intern Med. 2013 Apr 22;173(8):657-62; discussion 663. doi: 10.1001/jamainternmed.2013.351. PMID 23529201
- [Background] Tsafrir Z, Korianski J, Almog B, Many A, Wiesel O, Levin I. Effects of Fatigue on Residents' Performance in Laparoscopy. J Am Coll Surg. 2015 Aug;221(2):564-70.e3. doi: 10.1016/j.jamcollsurg.2015.02.024. Epub 2015 Mar 4. PMID 26081177
- [Background] Huffmyer JL, Moncrief M, Tashjian JA, Kleiman AM, Scalzo DC, Cox DJ, Nemergut EC. Driving Performance of Residents after Six Consecutive Overnight Work Shifts. Anesthesiology. 2016 Jun;124(6):1396-403. doi: 10.1097/ALN.0000000000001104. PMID 27028468
- [Background] Landrigan CP, Rothschild JM, Cronin JW, Kaushal R, Burdick E, Katz JT, Lilly CM, Stone PH, Lockley SW, Bates DW, Czeisler CA. Effect of reducing interns' work hours on serious medical errors in intensive care units. N Engl J Med. 2004 Oct 28;351(18):1838-48. doi: 10.1056/NEJMoa041406. PMID 15509817
- [Background] Barger LK, Cade BE, Ayas NT, Cronin JW, Rosner B, Speizer FE, Czeisler CA; Harvard Work Hours, Health, and Safety Group. Extended work shifts and the risk of motor vehicle crashes among interns. N Engl J Med. 2005 Jan 13;352(2):125-34. doi: 10.1056/NEJMoa041401. PMID 15647575
- [Background] Ayas NT, Barger LK, Cade BE, Hashimoto DM, Rosner B, Cronin JW, Speizer FE, Czeisler CA. Extended work duration and the risk of self-reported percutaneous injuries in interns. JAMA. 2006 Sep 6;296(9):1055-62. doi: 10.1001/jama.296.9.1055. PMID 16954484
- [Background] Goldstein MJ, Kim E, Widmann WD, Hardy MA. A 360 degrees evaluation of a night-float system for general surgery: a response to mandated work-hours reduction. Curr Surg. 2004 Sep-Oct;61(5):445-51. doi: 10.1016/j.cursur.2004.03.013. PMID 15475093
- [Background] Ko JS, Readal N, Ball MW, Han M, Pierorazio PM. Call Schedule and Sleep Patterns of Urology Residents Following the 2011 ACGME Reforms. Urol Pract. 2016 Mar;3(2):147-152. doi: 10.1016/j.urpr.2015.05.011. PMID 27840844
- [Background] Reed DA, Fletcher KE, Arora VM. Systematic review: association of shift length, protected sleep time, and night float with patient care, residents' health, and education. Ann Intern Med. 2010 Dec 21;153(12):829-42. doi: 10.7326/0003-4819-153-12-201012210-00010. PMID 21173417
- [Background] Wang Y, Loparo KA, Kelly MR, Kaplan RF. Evaluation of an automated single-channel sleep staging algorithm. Nat Sci Sleep. 2015 Sep 18;7:101-11. doi: 10.2147/NSS.S77888. eCollection 2015. PMID 26425109